CLINICAL TRIAL: NCT04938375
Title: Safety Profile of the Combination of Levosimendan and IV Beta Blocker in Cardiogenic Shock: a Retrospective Study
Acronym: SeLeBêta
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Sponsor
Other Study IDs: 2021PI069
Record Dates: First submitted 2021-06-17; First posted 2021-06-24 (Actual); Last update posted 2021-06-24 (Actual); Status verified 2021-06

CONDITIONS: Cardiogenic Shock; Arrythmia
MeSH Terms: conditions — Shock, Cardiogenic; Arrhythmias, Cardiac

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this study is to assess the safety profile of the combination of Levosimendan and beta blocker in cardiogenic shock with arrythmia.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients admitted to the ICU for cardiogenic shock who received esmolol or landiolol within 7 days of a levosimendan treatment

Exclusion Criteria:

* Patient's opposition

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients admitted to the ICU for cardiogenic shock who received esmolol or landiolol within 7 days of a levosimendan treatment
Sampling Method: Non-Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2016-01-01 (Actual); Primary Completion 2021-06-30 (Estimated); Study Completion 2021-07-30 (Estimated)

PRIMARY OUTCOMES:
To record adverse events and observe the safety profile of patients in cardiogenic shock who received concomitant treatment with Levosimendan and IV beta blocker | From the start of the beta blocker until 7 days after the start of the Levosimendan treatment
  Incidence of adverse events leading to discontinuation of beta blocker: bradycardia/high-grade atrioventricular block/hypotension/noradrenaline increase/crystalloid resuscitation

SECONDARY OUTCOMES:
Measure cardiac rhythm control; Measure heart rate control; Measure beta blocker dosages administered without adverse effects; Measure veno-arterial extra corporeal membranous oxygenation weaning rate; Measure resuscitation mortality | From the start of the beta blocker until 7 days after the start of the Levosimendan treatment ; Haemodynamic changes will be recorded every 2 hours from the start of the beta blocker
  Description of adverse events related to beta blocker Efficacy of beta blocker (rhythm and/or rate control) Time to resolution after discontinuation of beta blocker in case of adverse event Maximum dosage of well-tolerated beta blocker; Evolution of the haemodynamic profile in the hours following the introduction of the beta blocker Resuscitation mortality Weaning from veno-arterial ECMO at D7 of Levosimendan treatment